CLINICAL TRIAL: NCT01794429
Title: Treatment of Antipsychotic-associated Obesity With a GLP-1 Analogue
Acronym: TAO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bjorn H. Ebdrup (Other)
Responsible Party: Sponsor-Investigator, Bjorn H. Ebdrup, MD PHD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT nr: 2012-005404-17
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Metabolic Syndrome X; Drug-induced Obesity; Schizophrenia
Keywords: Obesity; The Metabolic Syndrome/disturbances; Drug-induced adipositas; Schizophrenia; GLP-1 analogue; cerebral effects
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Schizophrenia | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subcutaneum injection of placebo once-weekly for 3 months
  Interventions: Drug: Placebo
- exenatide (Active Comparator): Subcutaneum injection of exenatide once-weekly for 3 months
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Subcutaneum injection of exenatide once-weekly for 3 months
  Other Names: Bydureon
  Arms: exenatide
Drug: Placebo — Subcutaneum injection of placebo once-weekly for 3 months
  Arms: Placebo

SUMMARY:
To examine if 3 months of treatment with a GLP-1 (glucagon-like-peptide-1) analogue can induce weight loss in obese, non-diabetic patients with a diagnosis within the schizophrenic spectrum.

The investigators will also examine possible associations between GLP-1 treatment and peripheral metabolic parameters such as change in body fat and HbA1c. Moreover, the GLP-1 analogue treatment will be associated with the effects/changes on cognition and subjective quality of life. Possible cerebral effects (pro-cognitive) of the GLP-1 analogue treatment will associated and correlated with changes in the brain, functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
The primary endpoint is weight loss after 3 months of treatment with the GLP-1 analogue exenatide (Bydureon®).

Secondary endpoints comprise both physiological/metabolic parameters and cognitive measurements:

* Metabolic endpoints include amongst others: changes in body fat (DEXA-scan) and changes of the HbA1c(average blood glucose levels), cholesterol and triglycerides. Moreover physiological effects will be examined eg possible effect on central/peripheral bloodpressure and heart rate.
* Cerebral endpoints will be investigated via functional magnetic resonance imaging (fMRI); including potential neuroprotective effects of exenatide. The main focus is potential hippocampal volume changes and potential changes in cerebral blood flow. Functional MRI will provide this data and the images will be correlated to both cognitive tests and questionnaires.
* Cognitive endpoints comprise potential improvements in cognition with focus on specific memory tests (BACS, DART and Rey's Complex Figure) and possible improvements in subjective quality of life (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years
* Diagnosis of the schizophrenia spectrum (ICD-10: F20.x, F25.x)both in-patients and out-patients will be included
* Current and unchanged treatment with at least one antipsychotic drug (FGA and/or SGA and/or depot treatment)
* BMI ≥30 kg/m2
* HbA1c < 6,5 %

Exclusion Criteria:

* Substance dependence (ICD-10: F1x.2 (apart from nicotine addiction F17.2))
* Diabetes or HbA1c ≥6.5%
* Contraindications to MRI (metal implants, pacemakers, severe claustrophobia, ≥150 kg (max. bed weight in the MRI scanner))
* Previous head trauma with a loss of consciousness for more than 5 minutes
* Pregnancy (screened by urine human chorionic gonadotropin (hCG),lactation or no acceptance to use effective contraception during the intervention period
* Severe somatic disease, including inflammatory bowel disease and chronic ketoacidosis
* Allergy to exenatide
* Coercive measures according the Danish Law of Psychiatry
* conditions that according to sponsor are not congruous with participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months
  The primary endpoint is weight loss after 3 months of treatment with a GLP-1 analogue.

SECONDARY OUTCOMES:
Effects of GLP-1-analogue treatment on body fat composition | 3 months
  The investigators will explore potential effects of GLP-1 analogue treatment on different peripheral metabolic parameters: mainly changes in body fat composition (measured by DEXA-scan) and effects on HbA1c, triglycerides and cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Pelle L Ishøy, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Cnsr/Cins, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Ishoy PL, Fagerlund B, Broberg BV, Bak N, Knop FK, Glenthoj BY, Ebdrup BH. No cognitive-enhancing effect of GLP-1 receptor agonism in antipsychotic-treated, obese patients with schizophrenia. Acta Psychiatr Scand. 2017 Jul;136(1):52-62. doi: 10.1111/acps.12711. Epub 2017 Mar 5. PMID 28260235
- [Derived] Ishoy PL, Knop FK, Broberg BV, Bak N, Andersen UB, Jorgensen NR, Holst JJ, Glenthoj BY, Ebdrup BH. Effect of GLP-1 receptor agonist treatment on body weight in obese antipsychotic-treated patients with schizophrenia: a randomized, placebo-controlled trial. Diabetes Obes Metab. 2017 Feb;19(2):162-171. doi: 10.1111/dom.12795. Epub 2016 Nov 14. PMID 27717222
- [Derived] Ishoy PL, Knop FK, Broberg BV, Baandrup L, Fagerlund B, Jorgensen NR, Andersen UB, Rostrup E, Glenthoj BY, Ebdrup BH. Treatment of antipsychotic-associated obesity with a GLP-1 receptor agonist--protocol for an investigator-initiated prospective, randomised, placebo-controlled, double-blinded intervention study: the TAO study protocol. BMJ Open. 2014 Jan 8;4(1):e004158. doi: 10.1136/bmjopen-2013-004158. PMID 24401727